CLINICAL TRIAL: NCT01057368
Title: The Effects of Well-being Interventions on Affect, Attention, Sleep, Social Stress and Pain Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: WBP01-AT004952; P01AT004952 (NIH)
Record Dates: First submitted 2010-01-22; First posted 2010-01-27 (Estimated); Last update posted 2014-06-05 (Estimated); Status verified 2014-06

CONDITIONS: Health; Mental Health
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Mindfulness Based Stress Reduction (Active Comparator)
  Interventions: Behavioral: Mindfulness Based Stress Reduction (MBSR)
- Health Enhancement Program (Active Comparator)
  Interventions: Behavioral: Health Enhancement Program (HEP)
- Wait List Controls (No Intervention)
- Long Term Meditators (Active Comparator)
  Interventions: Behavioral: Day of intensive meditation practice

INTERVENTIONS:
Behavioral: Day of intensive meditation practice — Long-term meditators practice for ~6 hours of meditation at each time point
  Arms: Long Term Meditators
Behavioral: Mindfulness Based Stress Reduction (MBSR) — 8-week class designed to enhance well-being through training in mindfulness meditation
  Other Names: MBSR
  Arms: Mindfulness Based Stress Reduction
Behavioral: Health Enhancement Program (HEP) — 8-week class designed to enhance well-being through training in physical activity, functional movement, music therapy, and nutrition
  Other Names: HEP
  Arms: Health Enhancement Program

SUMMARY:
This study is focused on the brain mechanisms and peripheral biological correlates of two different forms of meditation--mindfulness-based and compassion/loving-kindness. Project 1 is focused on the impact of compassion/loving-kindness meditation on emotional reactivity and emotion regulation. Project 2 is focused on the neural and behavioral correlates of mindfulness meditation and attention and pain regulation. In addition, Project 2 will examine the relations between changes in oscillatory rhythms during meditation and attention and pain processing. Project 3 will examine the impact of meditation on spontaneous brain activity during sleep. This project will also examine the impact of intensive meditation on regional changes in slow wave activity during subsequent sleep. Each of these projects will be conducted on the same participants so that interrelations among the various measures collected in the different projects can be examined. We believe that this study will dramatically advance the understanding of the mechanisms by which meditation produces changes in behavioral and biological processes.

ELIGIBILITY:
Inclusion Criteria:

* MRI safe

Exclusion Criteria:

* Not available for scheduled visits or applicable interventions
* Current medical conditions that may affect outcome measures, including chronic inflammatory diseases, asthma, serious mental health diagnoses, chronic pain conditions, a personal history of seizures
* Regularly taking medications that may affect outcome measures, including pain medications, corticosteroids, immuno-suppressants, prescription sleep medications, psychotropic medications
* Alcohol or non-prescription drug problems
* Night-shift worker
* Diagnosed sleep disorder or habits, such as late bedtime, that would prevent enough sleep in the laboratory
* Previous training related to one of the two active interventions for meditation naive participants
* Unwillingness or inability to engage in intervention activities as determined by participant or their primary care physician
* Currently pregnant or planning on becoming pregnant in the next year
* Currently nursing
* Current IUD

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
MRI BOLD | Pre, Post, Follow-up (WL & LTP)
EEG | Pre, post, & follow-up (WL & LTP)
Salivary Cortisol | Pre, post, & follow-up (WL & LTP)
Behavioral | Pre, post, & follow-up (WL & LTP)
Self-report | Pre, post, & follow-up (WL & LTP)

SECONDARY OUTCOMES:
Self-report | Pre, post, & follow-up (WL & LTP)

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Davidson, PhD, Principal Investigator — UW-Madison
Locations (3):
- United States (3):
  - The Wisconsin Sleep Laboratory, Madison, Wisconsin
  - UW-Health Sports Medicine & Integrative Medicine Program, Madison, Wisconsin
  - UW-Madison, Laboratory for Affective Neuroscience, Madison, Wisconsin

REFERENCES:
- [Derived] Wielgosz J, Kral TRA, Perlman DM, Mumford JA, Wager TD, Lutz A, Davidson RJ. Neural Signatures of Pain Modulation in Short-Term and Long-Term Mindfulness Training: A Randomized Active-Control Trial. Am J Psychiatry. 2022 Oct;179(10):758-767. doi: 10.1176/appi.ajp.21020145. Epub 2022 Jul 28. PMID 35899379